CLINICAL TRIAL: NCT02241707
Title: Does Minimal Post-operative Compression Affect the Outcome for Endovenous Ablation in Treating Varicose Vein Patients?
Status: Withdrawn | Type: Observational
Why Stopped: Since reorganization of the institute, this study is aborted. No patient was recruited.
Sponsor: NYC Surgical Associates (Other)
Responsible Party: Sponsor
Other Study IDs: NYCSA-2014-01
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Varicose Vein; Venous Insufficiency
Keywords: Varicose vein; Endovenous ablation; Compression
MeSH Terms: conditions — Varicose Veins; Venous Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
In this proposal, the investigators seek to determine whether a reduced compression after endovenous ablation procedure in treating superficial venous insufficiency affects the outcomes. This study involves only the use of the compression stocking post endovenous ablation procedure and everything else is standard according to current guidelines.

The investigators general strategy will be to determine the role of a minimal post-operative compression and the status of patient satisfaction including (1) Success closure rate of the treated vein. (2) Less pain; (3) Easier accepted by the patients.

DETAILED DESCRIPTION:
All adults with varicose vein who are here in the investigators clinic to seek for endovenous ablation treatments will be invited to participate in this study. The participation in this research is entirely voluntary.

A. Each patient is given a code number instead of ID(identification) in the chart. Eligible patients according to their vein size are divided into following groups using a computer-generated randomization list:

1. Vein diameter between 5.5 and 6.7 mm, Post-op compression 1 day;
2. Vein diameter between 5.5 and 6.7 mm, Post-op compression 7 days;
3. Vein diameter between 6.8 and 8.5 mm, Post-op compression 3 days;
4. Vein diameter between 6.8 and 8.5 mm, Post-op compression 7 days.

B. Researchers: Data collectors and ultrasound technicians are blinded to the type of intervention, using code instead of patient's ID. The operating surgeon will not be the one who collects data. Performing physicians master these endovenous procedure techniques equally, have performed a minimum of 20 procedures independently.

C. Device: Graduated medical compression hosiery, 15-20mmHg. BrightLife Direct, Washington, DC. Endovenous ablation device: 1. Radiofrequency Ablation- FDA approval 1999, VNUS RFG2, San Jose, CA; 2. Endovenous Laser ablation- FDA approval Jan 2002, TVS 1470 by Total Vein System. Wavelength 1470nm, Nano Laser System device, Houston, TX. These two procedures are standard care under current guideline.

D. The research takes place over 12 months in total. During that time, it will be necessary for each patient to come to the clinic 6 times, for 1 hour each. The investigators would like to meet with every patient 1 week and 1, 3, 6, 12 months after the procedure respectively for a check-up.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and older
2. Diagnosis - symptoms (pain, burning, itching, cramping, heaviness and tiredness of leg, restless leg, swelling leg, etc.) and clinical signs (dilated veins, lipodermatosclerosis, color and texture changes of the skin, edema of leg, wound) correlates with vein diameter >5.5mm and reflex (>0.5 sec) in the upright position identified with duplex ultrasound
3. Severity/ classification - CEAP(clinical, etiologic, anatomic, and pathophysiologic) 3 or higher
4. Fail to a minimum of three months of nonoperative management (leg elevation, avoidance of prolonged standing, weight reduction, daily exercise for 30 min, prescription strength gradient compression garments, NSAIDs<nonsteroidal antiinflammatory drug>)
5. Post endovenous ablation (VNUS or laser) of the great saphenous vein (GSV) or small saphenous vein (SSV).

Exclusion Criteria:

1. Documented allergy or intolerance to compression hosiery
2. Treated vein greater than 8.5 in diameters.
3. Previous history of DVT(deep venous thrombosis); Known prothrombotic state.
4. Arterial insufficiency as determined by ABI(ankle-brachial index)<0.5.
5. Obesity (BMI >35, class II).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults, both male/female, with varicose vein who are here in our clinic to seek for endovenous ablation treatments will be invited to participate in this study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Vein closure success rate. | up to 12 months.
  Vein closure success rate determined by clinical evidence of symptom improvement and post-procedure duplex ultrasound @ 7 days, 1, 3, 6, 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Huang, MD, Study Director — NYC Surgical Associates; David A Greuner, MD, Principal Investigator — NYC Surgical Associates
Locations (1):
- NYC Surgical Associates, 555 Passaic Ave, Suite 10, West Caldwell, New Jersey, United States